CLINICAL TRIAL: NCT05002504
Title: Craniosacral Therapy as a Neurodevelopmental Correction for the Improvement of Children's Balance and Coordination.
Brief Title: Craniosacral Therapy Children's, Balance-Coordination
Acronym: CS-CHILDREN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Principal Investigator, Clinica Gema Leon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ART-GLB-CS-EQUILIB-COORD
Record Dates: First submitted 2021-08-07; First posted 2021-08-12 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Healthy Children
Keywords: Balance; Coordination; Craniosacral therapy; infants; physiotherapy

STUDY DESIGN:
Intervention Model Description: 25 patients in the placebo group (group 1), 30 patients in the craniosacral therapy group (group 2) and 31 patients in the balance and coordination therapy group (group 3)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will not know whether they will be treated or given a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients receiving craniosacral therapy (Experimental): 30 children without previous pathology receiving craniosacral therapy
  Interventions: Diagnostic Test: A series of questions were asked to the children's parents in a virtual questionnaire; Diagnostic Test: neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI); Procedure: Therapy sessions
- Patients receiving balance and coordination therapy (Active Comparator): 31 patients without previous pathology receiving balance and coordination therapy
  Interventions: Diagnostic Test: A series of questions were asked to the children's parents in a virtual questionnaire; Diagnostic Test: neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI); Procedure: Therapy sessions
- Patients receiving placebo (Placebo Comparator): 25 patients without previous pathology receiving placebo
  Interventions: Diagnostic Test: A series of questions were asked to the children's parents in a virtual questionnaire; Diagnostic Test: neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI); Procedure: Therapy sessions

INTERVENTIONS:
Diagnostic Test: A series of questions were asked to the children's parents in a virtual questionnaire — A series of questions were asked to the children's parents in a virtual questionnaire on physical characteristics, previous health assessments and observations of their balance and coordination in front of their children
  Other Names: questions were asked to the children's parents
Diagnostic Test: neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI) — the school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which evaluates five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. The results are assigned in age-adjusted percentages, classified as: low (0-49%), normal (50-79%) and high (80-100%). Low and high values are considered impairments in one or more of the areas evaluated. Evaluation of the Battelle scale was carried out before and after the therapy sessions.
  Other Names: "Battelle Developmental Inventory" (BDI)
Procedure: Therapy sessions — Seven treatment sessions were carried out with the balance and coordination therapeutic exercise techniques (group 3) most frequently used for the treatment of these pathologies; seven sessions of craniosacral therapy (group 2) as corrective and preventive in possible alterations during infant neurodevelopment and finally seven sessions simulating craniosacral therapy on a placebo group (group 1) as a control of the treatments used.

SUMMARY:
Coordination and balance are manifested as motor skills or abilities that are acquired as the Central Nervous System develops. In the infant stage, these qualities help guide specialists to recognize possible abnormalities that at first glance seem banal, but that, as time goes by, acquire greater difficulty, causing even more complex problems in the long term. Craniosacral therapy could help these skills to be correctly established during growth, correcting such impairment in time during neurodevelopment. Objective: To correct possible alterations that occur during infant growth related to balance and coordination in neurodevelopment, by means of craniosacral therapy compared with the specific therapy of balance and coordination usually used in pathologies diagnosed of this caliber. Design: Longitudinal-experimental study with a population of 86 apparently healthy children. Setting/Participants: 86 children were treated without excluding sex and divided into three groups: placebo group (n=25), craniosacral therapy group (n=30) and balance and coordination therapy group (n=31). Interventions: group 1 (placebo), group 2 (craniosacral therapy) group 3 (balance and coordination therapy). Results: The Battelle scale prior to the therapies developed in the study showed balance and coordination imbalances in the participants of the three groups, with lower percentages in the placebo treatment. Sessions from the 2nd to the 7th of treatment show increasing percentages and fluctuating for craniosacral therapy between 51% to 56% and 100% satisfaction, significantly valued. As for balance and coordination therapy, satisfaction percentages are evident only in the 6th and 7th sessions, with statistically significant values. Finally, the Battelle post-therapy assessment scale shows a higher number of participants in the percentages classified as normal (50-80%) in the craniosacral therapy group, improving the evaluated parameters with statistically significant values. Conclusion: The study shows that craniosacral therapy can not only act as a treatment for the improvement of children's balance and coordination, but also helps small corrections during children's neurodevelopment, avoiding the evolution of pathologies in the long term. It is therefore necessary for a more prompt, total and lasting correction of these skills in the infant.

DETAILED DESCRIPTION:
Design:

A longitudinal-experimental study was carried out with a child population of 86 children aged 6 to 8 years old without excluding sex in a school group in Cordoba (Spain).

Participants:

Eighty-six apparently healthy children between 6 and 8 years of age were treated as prevention in balance and coordination motor skills at the Gema León physiotherapy clinic in Córdoba (Spain). The children were divided into three groups: 25 patients in the placebo group (group 1), 30 patients in the craniosacral therapy group (group 2) and 31 patients in the balance and coordination therapy group (group 3).

Primary outcome: A series of questions were asked to the children's parents in a virtual questionnaire on physical characteristics, previous health assessments and observations of their balance and coordination in front of their children. On the other hand, the school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which evaluates five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. The results are assigned in age-adjusted percentages, classified as: low (0-49%), normal (50-79%) and high (80-100%). Low and high values are considered impairments in one or more of the areas evaluated.

Secondary outcome: Seven treatment sessions were carried out with the balance and coordination therapeutic exercise techniques (group 3) most frequently used for the treatment of these pathologies; seven sessions of craniosacral therapy (group 2) as corrective and preventive in possible alterations during infant neurodevelopment and finally seven sessions simulating craniosacral therapy on a placebo group (group 1) as a control of the treatments used.

The effectiveness values of the therapies were expressed as percentages of satisfaction with the classifications of 25 to 28% (apparent changes < to half of the sample in each therapy group), 51 to 56% (apparent changes in half of the sample in each therapy group) and 100% (apparent changes > to half of the sample in each therapy group). From the above, the absolute values of the sample in each therapy group are set as follows.

Data analysis:

The variables were expressed as mean, absolute and relative frequency. The chi-square test was used to analyze the differences between age ranges, balance and coordination problems versus physical therapy sessions performed, as well as the association between values of the Battelle scale of child neurodevelopment before and after the treatments. A confidence level of 95% was established, considering as statistically significant a value of p a value of p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* healthy children
* aged 6 to 8 years old
* school group

Exclusion Criteria:

* unhealthy children
* ages outside the 6-8 age range

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
"Series of questions to the children's parents" | two weeks
  A series of questions were asked to the children's parents in a virtual questionnaire on physical characteristics, previous health assessments and observations of their balance and coordination in front of their children
"Battelle Developmental Inventory" (BDI) | two weeks
  On the other hand, the school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which evaluates five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. The results are assigned in age-adjusted percentages, classified as: low (0-49%), normal (50-79%) and high (80-100%). Low and high values are considered impairments in one or more of the areas evaluated

SECONDARY OUTCOMES:
"Number of participants in each therapy group" | Seven weeks
  86 children were treated under stipulated physiotherapy techniques without excluding sex or age and divided into three groups: placebo group (n = 25), craniosacral therapy group (n = 30) and balance and coordination therapy group (n = 31). Each of the groups received the same number of therapeutic sessions (n = 7) spread over an equal period of time (one weekly session).
"The effectiveness values of the therapies for each group" | seven weeks
  The effectiveness values of the therapies were expressed as percentages of satisfaction with the classifications of 25 to 28% (apparent changes < to half of the sample in each therapy group), 51 to 56% (apparent changes in half of the sample in each therapy group) and 100% (apparent changes > to half of the sample in each therapy group).
"Pre-treatment Battelle Scale" | two weeks
  The pre-treatment assessments with the Battelle scale performed by the teachers evidenced the value of participants in all percentage ranges (low, normal and high), showing unevenness or alterations in primary explorations or assessments such as balance on two feet with eyes open and closed, on one foot with eyes open and closed (in neutral pelvis position), assessment of coordination in fast and slow movements and assessment of the coordination of the weaker side within their motor skills
"Post-treatment Battelle Scale" | two weeks
  The evaluation by the teachers with the Battelle scale after the treatment shows statistically significant values in the participants of the craniosacral therapy group (n=30), improving the parameters that they evaluate with respect to neurodevelopment, with 0% being in the low values (0-50) and 93% in normal values (50-80), rectifying the possible corrections made by means of this therapy
"percentages of satisfaction from 1st to the 7th therapy sessions" | seven weeks
  Significance values are observed for craniosacral therapy participants (n=30) showing apparent changes in gradual increases in the categories of 25-28% satisfaction from the 2nd session (n=20), moving to 51-56% satisfaction in the 3rd session (n=18) and swinging in gradual increases towards 100% satisfaction by the 5th session (n=15), showing that craniosacral therapy regulates small weaknesses or alterations previously observed during the balance and coordination exploration.
  During the sixth treatment session, craniosacral therapy shows higher percentages of apparent changes that position it with better satisfaction compared to balance and coordination therapy.
  The last treatment session presented a greater percentage advantage in the craniosacral therapy in relation to the balance and coordination therapy, ratifying the values previously exposed.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero Carmona, Study Chair — Universidad de Córdoba
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
The request for the data will be studied and considered upon prior and justified request.

REFERENCES:
- Available data/document: Clinical Study Report — http://dx.doi.org/10.1016/S0482-5985(05)74383-2 — Shapiro F, Forriol F. El cartílago de crecimiento: biología y biomecánica del desarrollo. Rev Ortop y Traumatol [Internet]. 2005;49(1):55-67.
- Available data/document: Clinical Study Report — http://dx.doi.org/10.1016/j.ft.2012.01.003 — Vázquez M, Rodríguez A, Arroyo A, Benjumea A. Desalineaciones de los miembros inferiores en niños con síndrome de Down. Fisioterapia [Internet]. 2012;34(4):140-5.
- Available data/document: Clinical Study Report — http://doi.org/10.1016/j.ft.2018.10.003 — Gatti C, Montero S. Effectiveness of treadmill training on gait development in children with Down syndrome: A systematic review. Fisioterapia [Internet]. 2019;41(1):37-47
- Available data/document: Clinical Study Report — http://scielo.sld.cu/scielo.php?script=sci%7B%5C_%7Darttext%7B%5C&%7Dpid=S0864-03002019000200086%7B%5C&%7Dlang=es%7B%5C%25%7D0Ahttp://scielo.sld.cu/pdf/ibi/v38n2/1561-3011-ibi-38-02-86.pdf — Taboada J, Díaz L, Hernández M. Restauración del patrón biomecánico de la marcha en niños cubanos. Rev Cuba Investig Biomédicas [Internet]. 2019;38(2):86-103
- Available data/document: Clinical Study Report — http://doi.org/10.1016/j.ft.2018.10.001 — Millar P, Navarro J, Martella D, Gallardo C. Prevalencia de alteraciones del neurodesarrollo motriz en niños prematuros sin diagnóstico de parálisis cerebral. Fisioterapia [Internet]. 2018;40(6):305-11.
- Available data/document: Clinical Study Report — http://dx.doi.org/10.1016/S1762-827X(14)68508-4 — Darmana R, Cahuzac J. Trastornos estáticos de los miembros inferiores y sus consecuencias sobre la marcha del niño. Trastornos rotacionales. EMC - Podol [Internet]. 2014;16(3):1-10.